CLINICAL TRIAL: NCT00919555
Title: Phase IIA Trial: Tretinoin and Pioglitazone HCL Combination Therapy in Amyotrophic Lateral Sclerosis
Brief Title: Combination Therapy in Amyotrophic Lateral Sclerosis (ALS)
Acronym: PNA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phoenix Neurological Associates, LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20071808
Record Dates: First submitted 2009-06-08; First posted 2009-06-12 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS Treatment; Tretinoin; Pioglitazone HCL; Actos; Tau levels; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Pioglitazone; Tretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tretionoin and Pioglitazone HCL (Active Comparator): 20 patients will be randomized blindedly to Tretinoin and Pioglitazone HCL
  Interventions: Drug: Pioglitazone and Tretinoin; Drug: Tretinoin and Pioglitazone HCL
- Sugar Pill (Placebo Comparator): 10 Patients will randomly receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone and Tretinoin — Tretinoin: 1 pill twice a day (10 mg/bid) Pioglitazone HCL: 1 pill once a day (30 mg/qd)
  Arms: Tretionoin and Pioglitazone HCL
Drug: Tretinoin and Pioglitazone HCL — Tretinoin 10 mg 1 pill po twice a day Pioglitazone HCL 30 mg 1 pill po once a day
  Arms: Tretionoin and Pioglitazone HCL
Drug: Placebo — Placebo
  Arms: Sugar Pill

SUMMARY:
The purpose of the study is to determine the safety and the efficacy of Tretinoin and Pioglitazone HCL in patients with ALS who are currently on Riluzole.

DETAILED DESCRIPTION:
Physicians at Phoenix Neurological Associates (PNA) are looking for individuals diagnosed with ALS to participate in a double-blind, placebo controlled study of Tretinoin and Pioglitazone HCL, used in combination with Riluzole, for treating ALS. This investigator initiated trial conducted by Dr. Todd Levine and Dr. David Saperstein will help determine whether Tretinoin and Pioglitazone HCL, in combination, can slow the progression of ALS.

At present, there is little to no effective therapy for ALS, nor is there a known cause. Therefore there is a tremendous unmet need for more effective therapy for this disease and that is why the physicians at PNA have been very interested in the role of developing a more active anti-excitotoxic cocktail for patients with ALS. Since recent data have suggested that inflammatory mechanisms may interact with and promote neurodegeneration (where cells in the spinal cord and brain are lost), there have been a number of anti-inflammatory treatment strategies that have been evaluated in animal models. Some studies have shown that mice that were given Pioglitazone HCL demonstrated improved muscle strength and body weight, exhibited a delayed disease onset as well as had a longer survival rate compared to non treated mice.

In addition to these studies, retinoic acids have been studied extensively in various models of the injured nervous system. These studies have shown that retinoic acids, such as Tretinoin may be neuroprotective and support axonal growth, which could in turn slow disease progression.

The purpose of this study is to determine if such a drug "cocktail" could offer the best chance of attaining a significant reduction in disease progression by utilizing currently available FDA-approved agents

ELIGIBILITY:
Inclusion Criteria:

* El Escorial Classification of laboratory supported probable, probable, or definite ALS
* Age 18 - 85 years
* Male or female
* FVC greater than or equal to 70% predicted

Exclusion Criteria:

* Patients with FVC below 1.5 L or below 70% predicted
* History of liver disease
* Severe renal failure (CrCl<30)
* History of coronary artery disease requiring placement of stents, bypass surgery or previous myocardial infarction
* EKG at baseline with evidence for previous myocardial infarction, cardiomyopathy, or arrhythmia
* History of intolerance to Riluzole, Tretinoin, or Pioglitazone HCL
* History of diabetes
* Any other comorbid condition which would make completion of trial unlikely

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Tretinoin and Pioglitazone HCL in patients with ALS | 3 years

SECONDARY OUTCOMES:
To determine if cerebrospinal fluid tau levels decline over the course of treatment and if the level of tau decline correlates with response in treatment measured by ALSFRS | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Levine, MD, Principal Investigator — Phoenix Neurological Associates, LTD
Locations (1):
- Phoenix Neurological Associates, LTD, Phoenix, Arizona, United States